CLINICAL TRIAL: NCT03872076
Title: Efficacy of a Protocol of Plyometric Exercises in the Improvement of Quadriceps Muscle Strength Versus Isometric Exercises With Theraband Elastic Band in Federated Water Polo Players. A Randomized Pilot Study.
Brief Title: Plyometric Exercises Versus Isometric Exercises With Theraband Elastic Band in Water Polo Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WATPLIO
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Muscle Loss
Keywords: Strengthening; Stability; Muscle Volume; Physical Effort; Randomized clinical trial
MeSH Terms: conditions — Muscular Atrophy | interventions — Plyometric Exercise; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric exercises (Experimental): The subjects included in the experimental group will carry out an intervention using plyometric exercises and isometric exercises with elastic band for the quadriceps muscle. Each session will last 15 minutes, taking place for 3 days a week, in a period of 8 weeks. The intervention will be made at the beginning of the training session.
  Interventions: Other: Experimental
- Isometric exercises (Active Comparator): The subjects included in the experimental group will carry out an intervention of isometric exercises with elastic bands for the quadriceps muscle. Each session will last 8 minutes, taking place for 3 days a week, in a period of 8 weeks. The intervention will be made at the beginning of the training session.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The Drom Jump technique with the legs flexed will be performed with the patient standing in front of a bench 30 cm high by 100 cm wide. The physiotherapist will be placed lateral to the athlete. The subject will be asked to jump up from the box or bench, with the hip and knees in semi-reflexion, with his hands on his hip and he will be asked for an explosive jump, followed by a jump downwards falling the floor of the same way.
  The technique of lateral jumps on cones will be carried out by means of unipodal jumps, achieving a distance of 50 cm between cones. The physiotherapist will stand in front of the athlete. The subject will be asked to perform a lateral unipodal explosive jump by flexing the hip and knee.
  Other Names: Plyometric exercises
  Arms: Plyometric exercises
Other: Control — Elastic bands will be combined with isometric exercises in 3 sets of 10 repetitions each. The exercises they will perform are front squat. On the one hand, separating the legs at the height of the shoulders with hip and knee flexion, with the elastic band above the knees, maintaining the position 20 seconds.
  In the following exercise, with the elastic band on the ankle, in unipodal support at the same time that the contralateral limb is free of support, the hip will be flexed at 45º with full knee extension, requesting the athlete to keep the tension 20 seconds, performing 3 sets of 10 repetitions.
  Other Names: Isometric exercises
  Arms: Isometric exercises

SUMMARY:
Introduction: The improvement of strength affects muscle volume, dynamic stability and sports performance in water polo athletes. Plyometric exercises can improve biomechanics, performance and the most explosive actions during sports. The work done with elastic bands will increase the effectiveness and the resistance on the isometric exercises developed.

Objectives: To evaluate the effectiveness of plyometric exercises in the increase of quadriceps muscle strength, volume and stability dynamic in female athletic of water polo players from 18 to 25 years old.

Study Design: A randomized, multicentric, single-blind clinical study with a follow-up period.

Methodology: 25 water polo players will be recruited and randomly assigned to the two study groups: experimental (plyometric exercises plus isometric exercises with elastic bands) and control (isometric exercises with elastic bands). The intervention will last for 8 weeks, with 3 weekly sessions, of 15 minutes each. The study variables will be: strength (measured with the RM test), muscle volume (using anthropometry), and dynamic stability (through the SEBT test). The analysis of normality will be carried out with the Shapiro Wilk test. In case of homogeneity of the groups, we will use parametric tests: t-student test of repeated measures (difference between evaluations) and ANOVA of repeated means (intra and intersubject effect).

Expected Results: It is expected to observe improvement in muscle strength and quadriceps volume, as well as dynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Swimmers with more than 2 years of sports practice
* Age range of 18 to 25 years
* Currently participate in national championships.

Exclusion Criteria:

* Have some type of musculoskeletal injuries at the time of the study
* Not signed the informed consent document.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline maximum strength in quadriceps after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Researchers will use the 1RM test to measure maximum strength by trial and error, taking into account the nRM (number of repetitions) performing a repetition for each series without exceeding 15 maximum repetitions, or even be effective in less than 10 maximum repetitions increasing the load in each series progressively, depending on the abilities of the athletes. We will perform 5 minutes of light activities, then one minute of stretching, heating of eight repetitions to 50% of 1RM, followed by three repetitions at 70% of 1RM. After 5 minutes of the interval, the 1RM test will be performed. The weight will increase progressively 5kg, three to five times until the maximum RM. The assessment of quadriceps muscle strength will be assessed through the full squat exercise. The unit of measurement is the Kg, indicating a greater amount of Kg, a greater maximum force in quadriceps

SECONDARY OUTCOMES:
Change from baseline muscle volume in quadriceps after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A metric tape will be used as a measuring instrument to assess muscle volume of quadriceps. Once the segment to be assessed is identified, we will make the assessment with the athlete in standing position. A mark will be made on the upper edge of the patella, and another one at 10 centimeters in the same plane of movement, in caudal-cranial direction. The evaluation will be carried out by measuring the entire contour on the marked lines, thus defining the different perimeters. This test has the centimeter (cm) as the unit of measurement. The higher the score, the more muscle volume the subject reflects in the valued segment.
Change from baseline dynamic stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The evaluation of the dynamic stability will be carried out through the use of the Star Excursion Balance Test. With the patient in a standing position, squatting on a limb without support will be requested. On the ground, 8 lines will be marked with a separation between them of 45 degrees forming a star. Data will be obtained in different planes (anterior, anterolateral, medial, posteromedial, posterolateral and posterior). The athlete must establish a stable base at the point of support and keep it in all directions, while trying to touch the lines with the most distal part of the foot and return to the starting position. This scale has the centimeter as a unit of measurement: the higher the score in centimeters, the more dynamic stability the athlete presents.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain